CLINICAL TRIAL: NCT00659620
Title: Mesenchymal Stem Cell Transplantation in the Treatment of Chronic Allograft Nephropathy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fuzhou General Hospital (Other)
Responsible Party: FUZHOU GENERAL HOSPITAL, FUZHOU GENERAL HOSPITAL
Organization: Organ Transplant Institute, China (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: fuzhough0712; fuzhough0712
Record Dates: First submitted 2008-04-14; First posted 2008-04-16 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2008-04

CONDITIONS: Kidney Transplant; Chronic Allograft Nephropathy
Keywords: Kidney Transplant; Chronic Allograft Nephropathy; Mesenchymal Stem Cell infusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): transplantation of mesenchymal stem cell
  Interventions: Biological: mesenchymal stem cell

INTERVENTIONS:
Biological: mesenchymal stem cell — transplantation of mesenchymal stem cell
  Other Names: MMF FK506

SUMMARY:
Mesenchymal Stem Cell (MSC) have been shown to have immunosuppressive and repairing properties. the investigators will infuse expanded MSC into patients who develop Chronic Allograft Nephropathy. The purpose of this study is to find out MSC is more effective in preventing organ rejection and maintaining kidney function.

DETAILED DESCRIPTION:
Kidney transplantation is a common procedure in hospitals, but organ rejection and chronic nephrotoxicity are potential problems for the patient. Approximately ninety percent of the protocol biopsies of renal allografts, performed at 18 months post transplantation, show histological lesions of chronic calcineurin nephrotoxicity. Mesenchymal Stem Cell (MSC) has been shown to have immunosuppressive and repairing properties. Some patient in this study will also receive two infusions of expanded MSC. This study will evaluate the safety and effectiveness of MSC infusions in patients .

This study will last 2 years. Participants will be randomly assigned to receive either the full immunosuppressive therapy and MSC infusions (Group 1) or immunosuppressive therapy alone (Group 2). Patients will undergo MSC infusions at the start of the study on Day 0. One year post- infusions, patients will be evaluated. At Months 12 participants will undergo kidney biopsies. Blood collection will occur at regular intervals, Serum creatinine and the estimated creatinine clearance will be monthly recorded. The transplanted kidney function will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of a renal allograft, Male and female patients age 18 to 60 years of age.
* Ability to provide written informed consent.
* The serum creatinine form 176umol/L(2mg/ml) to 440umol/L(5mg/ml)
* Renal biopsy Criteria: chronic allograft nephropathy (Banff I-II).
* Immunosuppressant:CNI and MMF and Sirolimus
* Written informed consent, compliant with local regulations.

Exclusion Criteria:

* Recipients with leucopenia (WBC < 3000/mm³), thrombocytopenia (Thr < 100.000/mm³),or hyperlipidemia (Tot Chol > 300 mg/dl or Triglycerides > 300 mg/dl).
* Recipients of multiple organs.
* Pregnant women.
* Previous history of malignancy
* Active infection including hepatitis B, hepatitis C, HIV, or TB as determined by a positive skin test or clinical presentation, or under treatment for suspected TB.
* Evidence of cardiovascular disease, existing congestive cardiac failure on physical exam and/or acute coronary syndrome in past 6 months.
* Inadequate compliance to treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2008-05; Primary Completion 2008-05 (Estimated); Study Completion 2010-05 (Estimated)

PRIMARY OUTCOMES:
Creatinine and creatinine clearance rate | 5

SECONDARY OUTCOMES:
Patient and graft survival [ Time Frame: At 1 years post-transplant ]. | 5
The proportion of renal biopsy after 12 months | 2
The incidence of infectious complications | 5
Incidence of adverse events associated with MSC and immunosuppression | 5

CONTACTS AND LOCATIONS:
Overall Officials: Jianming Tan T Jianming, professor, Principal Investigator — Fuzhou General Hospital
Locations (1):
- Fuzhou General Hospital, Fuzhou, Fujian, China